CLINICAL TRIAL: NCT02730819
Title: An Open-Label Pilot Study Evaluating the Effectiveness and Tolerability of a Topical Composition Therapy (2013-MCN-333) for the Treatment of Melasma
Brief Title: Topical Composition Therapy (2013-MCN-333) for the Treatment of Melasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jason Sluzevich, Assistant Professor of Dermatology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-005615
Record Dates: First submitted 2016-03-29; First posted 2016-04-07 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Illuminate Cream (Experimental): Illuminate Cream is a skin-lightening formulation containing multiple drugs, including a retinoid, calcineurin inhibitor, anti-tyrosinase agent and sunscreen microfine zinc oxide. Approximately 0.5 grams to be applied topically to affected areas of skin once per day for 20 weeks.
  Interventions: Drug: Illuminate Cream

INTERVENTIONS:
Drug: Illuminate Cream — Topical compound applied daily
  Other Names: 2013-MCN-333

SUMMARY:
The purpose of this research study is to gather information on the effectiveness and tolerability of a novel composition of existing U.S. Food and Drug Administration (FDA) approved topical medications for the treatment of moderate to severe melasma.

DETAILED DESCRIPTION:
Subjects with moderate to severe melasma will apply 0.5 grams (pea-sized) amount of Illuminate Cream topically to affected areas for 20 weeks. The change in Melasma Area and Severity Index (MASI) score will be evaluated a baseline and Weeks 4, 12, and 20.

The MASI score is a validated test, calculated by subjective assessment of 3 factors: Area (A) of involvement, Darkness (D), and Homogeneity (H), with the forehead, right malar region, left malar region, and chin, corresponding to 30%, 30%, 30% and 10% of the total face, respectively. The area of involvement in each of these 4 areas is given a numeric value of 0 to 6 (0 = no involvement; 1 = <10%; 2 = 10%-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; and 6 = 90-100%).

Darkness and homogeneity are rated on a scale from 0 to 4 (0 = absent; 1 = slight; 2 = mild; 3 = marked; and 4 = maximum). The score is calculated by adding the sum of the severity ratings for darkness and homogeneity, multiplied by the value of the area of involvement, for each of the 4 facial areas.

ELIGIBILITY:
Inclusion Criteria:

* Informed subject consent will be obtained from those patients meeting the following inclusion criteria:
* Male and female patients 18 to 65 years age
* Moderate to severe melasma, as measured by the Melasma Area Severity Index score greater than or equal to 16
* No prior use of topical skin-lightening agents for 1 month prior to study entry
* Good general health as confirmed by medical history
* Female patients of child-bearing potential with a negative urine pregnancy test who agree to use effective methods of birth control or remain abstinent during treatment. Participants must use birth control for the entire study and for at least 1 week after the last application of the study formulation. Acceptable methods of birth control include ongoing hormonal contraception methods, (such as birth control pills, patches, injections, vaginal ring, or implants), barrier methods (such as a condom or diaphragm used with a spermicide), intrauterine devices, tubal ligation, or abstinence
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol; and
* Patients who read and sign an approved informed consent for this study

Exclusion Criteria:

* Vulnerable study population
* Exposure to topical skin-lightening agents within 1 month of study entry, including:

  1. Topical corticosteroids
  2. Topical bleaching products
  3. Topical retinoids
* Use of systemic preparations within 1 month of study entry, including:

  1. Systemic corticosteroids
  2. Systemic cyclosporine, interferon
  3. Systemic acitretin, etretinate, isotretinoin
  4. Systemic methotrexate
  5. Systemic photoallergic, phototoxic and/or photosensitizing drugs
* UV light therapy and sunbathing
* Inability to communicate or cooperate with the Principal Investigator and/or Investigators due to language problems, poor mental development or impaired cerebral function
* Pregnant or nursing women
* Women planning a pregnancy within the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Sluzevich, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen at the Mayo Clinic in Jacksonville, Florida between May 2016 and September 2016 were enrolled in the study.
Period: Overall Study
Arm/Group | Illuminate Cream
Started | 19
Follow-up Week 2 | 15
Follow-up Week 4 | 16
Follow-up Week 8 | 14
Follow-up Week 12 | 11
Follow-up Week 16 | 11
Follow-up Week 20 | 10
Completed | 10
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Population: 19 participants were enrolled, but 3 did not return for any of the follow-up visits and were not included in any of the analyses.
Arm/Group | Illuminate Cream
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 38 [31 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color.
  Type I (scores 0-6) always burns, never tans Type II (scores 7-13) usually burns, tans minimally Type III (scores 14-20) sometimes mild burn, tans uniformly Type IV (scores 21-27) burns minimally, always tans well Type V (scores 28-34) very rarely burns, tans very easily Type VI (scores 35-36) Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Type 1 | 0
    Type 2 | 8
    Type 3 | 5
    Type 4 | 1
    Type 5 | 2
Use oral contraceptives [Count of Participants; unit: Participants] | 3
Use sunscreen daily [Count of Participants; unit: Participants] | 11
Melasma started with pregnancy [Count of Participants; unit: Participants] | 5
Received prior treatments for melasma [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Melasma Area and Severity Index (MASI) Score
Description: Severity of melasma in each of the four regions (forehead, right malar region, left malar region and chin) is assessed on % of the total area involved (A), darkness (D), and homogeneity (H).
  Scoring for % area involved: 0=none; 1=<10%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; and 6=90-100%. Darkness scoring (hyperpigmentation): 0=normal skin; 1=barely visible; 2=mild; 3=moderate; 4=severe. Homogeneity scoring: 0=normal skin color; 1=specks of involvement; 2=small patchy areas of involvement <1.5 cm diameter; 3=patches of involvement >2 cm diameter; 4=uniform skin involvement without any clear areas).
  To calculate the MASI score, the sum of the severity grade for darkness (D) and homogeneity (H) is multiplied by the numerical value of the areas (A) involved and by the percentages of the four facial areas (10-30%). Total MASI score: Forehead 0.3 (D+H)A + right malar 0.3 (D+H)A + left malar 0.3 (D+H)A + chin 0.1 (D+H)A. The total score can range from 0 (normal) to 48 (severe).
Time Frame: Baseline, 20 weeks
Population: 19 participants were enrolled, but 9 participants were lost to follow-up over the course of the study.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Illuminate Cream
Number analyzed (Participants) | 10
units on a scale | -11.4 [-15.3 to -3.6]
Statistical Analysis 1: Comparison: Illuminate Cream; P-values of 0.05 or lower were considered statistically significant; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Melasma Quality of Life Scale (MELASQOL)
Description: The Melasma Quality of Life Scale has 10 items, with responses ranging from 0 (no response) to 7 (bothered all the time. The range of possible scores is 0-70, with a higher score indicating a worse melasma-related quality of life.
Time Frame: baseline, 20 weeks
Population: 19 participants were enrolled, but 9 participants were lost to follow-up over the course of the study.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Illuminate Cream
Number analyzed (Participants) | 10
units on a scale | -10 [-35 to -1]
Statistical Analysis 1: Comparison: Illuminate Cream; P-values of 0.05 or lower were considered statistically significant; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Investigator Assessment of Global Improvement From Baseline
Description: The investigator compared the extent of melasma at 20 weeks to a full-face photograph obtained in a standardized manner at baseline. It is a dynamic 7-point scale (0=completely clear to 7=worse).
Time Frame: baseline, 20 weeks
Population: 19 participants were enrolled, but 9 participants were lost to follow-up over the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Illuminate Cream
Number analyzed (Participants) | 10
Participants
  0=Completely clear | 0
  1=Almost clear | 1
  2=Significant or marked improvement | 2
  3=Moderate improvement | 4
  4=Slight improvement | 3
  5=No change from baseline | 0
  6=Worse | 0

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Illuminate Cream
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Illuminate Cream (N=16)
Fell and broke ribs (Injury, poisoning and procedural complications) | 1 (1)
Peeling of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Irritation on face due to sun exposure (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 16 (20)
Scaling (Skin and subcutaneous tissue disorders) | 16 (30)
Dryness (Skin and subcutaneous tissue disorders) | 16 (40)
Stinging (Skin and subcutaneous tissue disorders) | 16 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes